CLINICAL TRIAL: NCT00409526
Title: Pilot Study: The Effect of Inhaled Iloprost on Oxygenation in Term and Near Term Infants With Pulmonary Hypertension. Testing Two Doses.
Brief Title: Inhaled Iloprost for the Treatment of Persistent Pulmonary Hypertension in the Term and Near Term Infants.
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Sub-Investigator left U of C
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14479B
Record Dates: First submitted 2006-12-07; First posted 2006-12-11 (Estimated); Last update posted 2014-06-02 (Estimated); Status verified 2014-05

CONDITIONS: Pulmonary Hypertension
Keywords: Iloprost; PPHN; Newborn; Pulmonary Hypertension; Term; Persistent Pulmonary Hypertension of the Newborn
MeSH Terms: conditions — Hypertension, Pulmonary; Persistent Fetal Circulation Syndrome | interventions — Iloprost

INTERVENTIONS:
Drug: Inhaled Iloprost — 50 micrograms for one hour followed by 100 micrograms for one hour
  Other Names: Ventavis

SUMMARY:
Inhaled Iloprost will be administered to near term infants with Persistent Pulmonary Hypertension of the Newborn in two different doses in order to test safety and efficacy in reducing pulmonary artery pressure.

DETAILED DESCRIPTION:
Infants eligible for the study will be divided into two arms according to oxygenation index: Infants in arm A (OI <20) will receive nebulized Iloprost in a lower dose (50 ng/kg/min) for one hour, and a higher dose (100 ng/kg/min) for another hour. Infants in arm B (OI>20) will receive NO, and in addition will receive nebulized Iloprost in a lower dose for one hour and a higher dose for another hour.

ELIGIBILITY:
Inclusion Criteria:

* Near-term infants (>34 gestational age) with evidence of persistent pulmonary hypertension and severe hypoxia(PaO2<100 mmHg with mechanical ventilation with FiO2=100%).

Exclusion Criteria:

* Major congenital malformation
* Congenital diaphragmatic hernia
* Structural cardiac anomalies
* Hydrops fetalis
* Pulmonary hemorrhage
* Severe perinatal depression
* Patients on high frequency oscillation ventilator

Max Age: 7 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1 (Actual)
Dates: Start 2006-12; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Oxygenation index and PaO2 after treatment with inhaled Iloprost. | three hours

CONTACTS AND LOCATIONS:
Overall Officials: Michael D Schreiber, MD, Principal Investigator — University of Chicago
Locations (2):
- Comer Children's Hospital, The University of Chicago Hospitals, Chicago, Illinois, United States
- Shaare Zedek Medical Center, Jerusalem, Israel